CLINICAL TRIAL: NCT01385215
Title: Strategies for Enhancing Mucosal Immunity to Influenza Vaccine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: John Sundy (Other)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00024277
Record Dates: First submitted 2011-04-25; First posted 2011-06-30 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Mucosal Immunity
Keywords: Vaccination; Mucosal Immunity; Nasal Immunization
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Fluzone
- Nasal Aerosol Immunization (Placebo Comparator)
  Interventions: Drug: Fluzone
- Nasal Droplet Immunization (Placebo Comparator)
  Interventions: Drug: Fluzone
- Intramuscular Immunization (Placebo Comparator)
  Interventions: Drug: Fluzone

INTERVENTIONS:
Drug: Fluzone — 0.5 ml/15 micrograms
  Arms: Intramuscular Immunization
Drug: Fluzone — 0.5 ml/60 micrograms
  Arms: Nasal Aerosol Immunization; Nasal Droplet Immunization; Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the influenza vaccine when administered nasally and intra-muscular (a "shot" of medicine given into a muscle). The investigators will measure the systemic (through out the body) and mucosal immune responses (how your body recognizes and defends itself against bacteria) to nasally administered influenza vaccine, and determine if nasal immunization results in immunity (your body's ability to avoid infections) within multiple mucosal compartments (ocular (eye), oral and reproductive), in comparison with intramuscular administration and placebo (inactive substance given in the same form as the active drug).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ages 18-50 years
* Non-smokers (defined as no tobacco use within the last 12 months and less than 10 pack-year lifetime tobacco use)
* Willing and able to provide written informed consent
* Able to speak and understand English
* Women of childbearing potential must have a negative serum pregnancy test.

Exclusion Criteria:

* Influenza vaccination within 6 months prior to screening date
* Symptoms of respiratory infection during the 14 days prior to screening
* Temperature >38.3o C during the period spanning 72 hours prior to screening and the time of immunization.
* History of allergy to egg, influenza vaccine or vaccine ingredients
* History of Guillain-Barre syndrome
* History of Bell's palsy
* Tonsillectomy, adenoidectomy or prior surgery to the paranasal sinus cavity.
* Physician diagnosis of or personal history of allergic or chronic rhinitis
* Physician diagnosis of or personal history of asthma
* Acute sinusitis within 30 days prior to screening
* Use of antibiotics within 14 days prior to screening
* Requirement for use of nasal corticosteroids for the period beginning 30 days prior to screening through final study visit
* Requirement for use of antihistamines (systemic, intranasal or intraocular) for the period beginning 72 hours prior to screening through final study visit
* Use of immunomodulating drugs or systemic corticosteroids within 6 months prior to screening (includes but is not limited to azathioprine, methotrexate, mycophenolate mofetil, tumor necrosis factor inhibitors, cyclosporine, tacrolimus)
* Past or present history of allergen immunotherapy to within the last 10 years.
* Students or employees who are under direct supervision by any of the investigators in this protocol are not eligible to participate.
* Subjects who abuse alcohol or illicit substances will be excluded.
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements.
* Nursing mothers.
* Other investigational medication use within 30 days of screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in hemagglutinin antibody titers from baseline to Day 28 in serum and mucosal secretions. | Baseline to Day 28
  Assessments will include hemagglutination inhibition and antibody isotypes determination.

SECONDARY OUTCOMES:
Number of subjects with adverse events. | Baseline to Day 28
Comparison of hemagglutinin antibody titers between intranasal and intramuscular route of administration, from baseline to Day 28. | Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: John Sundy, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States